CLINICAL TRIAL: NCT05257018
Title: A Phase II Study of R-CDOP Combined With Intrathecal Methotrexate for Diffuse Large B-cell Lymphoma Patients With High-risk of Central Nervous System Relapse
Brief Title: R-CDOP Combined With Intrathecal Methotrexate for DLBCL Patients With High-risk of CNS Relapse
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ji Dongmei, Associate Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DMS-LM-K001
Record Dates: First submitted 2021-12-20; First posted 2022-02-25 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Chemo-naive Diffuse Large B-cell Lymphoma; Doxorubicin Hydrochloride Liposome Injection; Methotrexate; Central Nervous System Relapsed; R-CDOP; Objective Response Rate; Progression Free Survival; 2-year CNS relapse rate
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- R-CDOP+intrathecal MTX (Experimental): R-CDOP+intrathecal MTX：
  * Rituximab 375 mg / m^2，D1
  * Cyclophosphamide 750 mg / m^2，D2
  * Doxorubicin Hydrochloride Liposome Injection 35mg / m^2，D2
  * Vincristine 1.4mg/m^2 (dose capped at 2 mg)，D2
  * Prednisone 50 mg， bid D2-6
  * Cycle1-5：Intrathecal MTX 12 mg + DXM 5 mg after chemotherapy （PK patients will be given 24h after chemotherapy）
  Interventions: Drug: R-CDOP+intrathecal MTX

INTERVENTIONS:
Drug: R-CDOP+intrathecal MTX — R-CDOP+intrathecal MTX：
  * Rituximab 375 mg / m^2，D1
  * Cyclophosphamide 750 mg / m^2，D2
  * Doxorubicin Hydrochloride Liposome Injection 35mg / m^2，D2
  * Vincristine 1.4mg/m^2 (dose capped at 2 mg)，D2
  * Prednisone 50 mg， bid D2-6
  * Cycle1-5：Intrathecal MTX 12 mg + DXM 5 mg after chemotherapy （PK patients will be given 24 h after chemotherapy）
  Other Names: Pegylated liposome doxorubicin（PLD）

SUMMARY:
This is a double-center, single-arm, phase 2 study to evaluate the efficacy and safety of R-CDOP regimen combined with intrathecal methotrexate in chemo-naive diffuse large B-cell lymphoma patients with high-risk of CNS relapse.

DETAILED DESCRIPTION:
Diffuse large B-cell lymphoma is the most common subtype of non-Hodgkin's lymphoma, accounting for 31% of all non-Hodgkin's lymphomas. At present, the standard treatment is R-CHOP (rituximab, cyclophosphamide, doxorubicin, vincristine, prednisone) Regimen. In DLBCL, central nervous system recurrence is rare, but once it occurs, it is often fatal. The prognosis of patients with central recurrence of DLBCL is very poor, and the median survival time is only 3.5-7 months.The CNS relapse rate of the R-CHOP regimen combined with MTX (methotrexate) intrathecal in high CNS-IPI DLBCL patients is approximately 12%.

This study was a phase II, prospective, single arm，double-center study, which requires a total of 83 DLBCL patients with high-risk of CNS relapse.

Patients will receive a total of 6-8 cycles of R-CDOP regimen, repeated every 3 weeks. Intrathecal MTX will be administered after the 1st-5th cycle of chemotherapy. All the patients will receive a mid-treatment PET scan after 4 cycles of chemotherapy. Patient achieves CR (complete response) after 4 cycles will continue to receive another 2 cycles of treatment. For those who achieve PR, another 4 cycles of chemotherapy will given.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 18 to 75 years;
2. ECOG performance status: 0-2;
3. Histopathologically confirmed untreated diffuse large B-cell lymphoma (cell origin can be distinguished according to Hans algorithm) , And fulfilled the following criteria for high-risk CNS recurrence:

   1. CNS-IPI 4-6;
   2. The lymphoma involved testis, breast (excluding unilateral breast and less than 5 cm mass), adrenal gland, kidney, paranasal sinus, paravertebral, and bone marrow and other sites;
   3. PCLBCL-leg;
4. Subjects have at least one measurable lesion: the long axis of the lymph node shall be>1.5 cm, the long axis of the extranodal lesions shall be>1.0 cm;
5. Bone marrow hematopoiesis was essentially normal: WBC≥3.5 ×10^9/L, ANC≥1.5×10^9/L, PLT≥80×10^9/L, Hb≥90 g/L. Abnormal peripheral blood indices, as a result of lymphoma invading the bone marrow or spleen, permitted enrollment at the discretion of the investigator;
6. Liver function: total bilirubin, ALT, AST < 1.5×UNL (upper limit of normal);
7. Renal function: Cr < 1.5×UNL and creatinine clearance≥30 ml/min;
8. Echocardiography or nuclide cardiac function testing with LVEF≥50%;
9. Patients in the reproductive period agreed to appropriate contraception. Women in the reproductive period had a negative serum pregnancy test within 2 weeks before enrollment;
10. Consent to provide pathological tissue specimens (wax blocks within half a year or 20 slides for paraffin tissue sections);
11. Life expectancy≥3 months;
12. Signed informed consent;

Exclusion Criteria:

1. Patients with a known history of severe allergy to humanized or murine mAbs, or any contraindication to R-CDOP, intrathecal MTX;
2. Patients with evidence of CNS involvement (baseline cerebrospinal fluid, imaging, symptoms);
3. Special types of diffuse large B-cell lymphoma patients who are not suitable for induction therapy with R-CDOP, such as PMBCL, double-hit large B-cell lymphoma, etc;
4. Clinically significant cardiac conditions, including severe cardiac insufficiency: New York Heart Association (NYHA) cardiac insufficiency class IV, unstable angina, acute myocardial infarction within 6 months prior to screening, congestive heart failure, and Q-Tc interval greater than 500 ms;
5. Those who had a second degree or greater operation within three weeks before treatment;
6. Diagnosed with a malignancy other than lymphoma or under treatment, with the following exceptions:

   1. Had received treatment with curative intent and had not developed malignancy with known active disease ≥ 5 years prior to enrollment;
   2. Basal cell carcinoma of the skin (other than melanoma) that has been adequately treated with no evidence of disease;
   3. Carcinoma in situ of the cervix that has been adequately treated with no evidence of disease;
7. Had significant coagulation abnormalities;
8. Any previous antilymphoma therapy other than short-term corticosteroids (up to 10 days);
9. Those with severe active infection;
10. Other serious, uncontrolled concomitant conditions that may affect protocol adherence or interfere with interpretation of results include uncontrolled diabetes mellitus, or pulmonary disease (interstitial pneumonia, obstructive pulmonary disease, and a history of symptomatic bronchospasm), hypertension, and others;
11. HBV (HBsAg positive and HBV-DNA ≥ 104 IU / ml), HCV (HCV antibody positive and HCV-RNA measurable); And subjects with other acquired, congenital immunodeficiency diseases, including but not limited to those with HIV infection;
12. Pregnant or lactating women;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2022-02-26 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
2-year central nervous system relapse rate | up to 6 years after the start of the study
  The proportion of patients with central nervous system recurrence within two years from enrollment accounted for all patients treated with drugs.
Concentration of doxorubicin in cerebrospinal fluid after using doxorubicin hydrochloride liposome injection | up to 4 years after the start of the study
  CSF doxorubicin concentrations 24 hours after the first 5 courses of lipso-doxorubicin infusion will be tested. Peak concentration of doxorubicin in CSF will be recorded, and the area under the curve will be calculated.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 years after enrollment of final patient
  Objective response rate measured as number of complete and partial response divided by the number of patients included.
2-year progression-free survival (PFS) rate | 2 years after enrollment of final patient
  Number of non-progression cases/all enrolled cases at 2 years
2-year event-free survival (EFS) rate | 2 years after enrollment of final patient
  Number of non-event cases/all enrolled cases at 2 years
Overall Survival (OS) | 2 years after enrollment of final patient
  Time from the date of enrollment to data of death from any cause, or date of lost follow-up, whichever comes first, and otherwise censored at time last known alive.
Adverse events | Since the signing of informed consent forms to 30 days after the last cycle
  Hematologic and non hematologic adverse event (CTCAE 4.03）
Cmax（maximum concentration） | Time from zero to Tmax
  The peak concentration of the drug
Tmax（maximum time） | Time from zero to Cmax
  The peak time of the drug
T1/2（drug half time） | The time it takes for blood concentration levels to drop by half
  The time it takes for blood concentration levels to drop by half
AUC（0-∞）（area under the curve） | Time from zero to ∞
  area under the concentration-time curve
AUC （0-t）（area under the curve from time zero to the last observation time | Time from zero to the last observation time
  area under the concentration-time curve from time zero to the time of last area area under the concentration-time curve from time zero to the last observation time

CONTACTS AND LOCATIONS:
Overall Officials: Dongmei Ji, doctor, Principal Investigator — Fudan University; Junning Cao, Doctor, Principal Investigator — Fudan University
Locations (2):
- China (2):
  - Dongmei Ji, Shanghai, Shanghai Municipality
  - Cancer Hospital affilicaited to Xinjiang Medical University, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: No